CLINICAL TRIAL: NCT02915952
Title: A Prospective, Non-blinded, Randomized Controlled Post-market Study Designed to Compare the Use of the Zip Surgical Skin Closure Device Versus Sutures for Skin Closure in Subjects Who Undergo a Cesarean Section Procedure.
Brief Title: Zip Incision Approximation vs. Suture for C-Section
Acronym: ZIPS-C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZipLine Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZipsC-006
Record Dates: First submitted 2016-09-16; First posted 2016-09-27 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: C.Surgical Procedure; Dehiscence, Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zip Closure Device (Active Comparator): The Zip device is a non-invasive, single use, sterile medical device for closure of the skin layer for surgical incisions or laceration repair.
  Interventions: Device: Zip Surgical Skin Closure Device
- Conventional Sutures (Active Comparator): Conventional subdermal (subcuticular) absorbable sutures
  Interventions: Other: Conventional Sutures

INTERVENTIONS:
Device: Zip Surgical Skin Closure Device — The Zip Surgical Skin Closure Device will be used for surgical wound closure in C-Section Surgery
  Other Names: Zip
  Arms: Zip Closure Device
Other: Conventional Sutures — Conventional Sutures will be used for surgical wound closure in C-Section Surgery
  Arms: Conventional Sutures

SUMMARY:
The study will evaluate the ZipLine Medical Surgical Skin Closure device (Zip)versus sutures when utilized for skin layer closure during wound closure of Cesarean Section Procedure.

DETAILED DESCRIPTION:
Cesarean-section birth is a very invasive surgical procedure. While the desired outcome focuses primarily on the successful delivery of a healthy baby and maintenance of the mother's health, the surgery involves a complex surgical closure process, starting with the uterus, and progressing through several layers of traditionally suture closure in several tissue planes. A successful closure results in no surgical site complications, with good patient comfort and a minimal scar being a desired outcome.

Conventional skin closure methods such as sutures are effective but have drawbacks. It has been suggested that the ideal method of wound / incision closure should be:

* fast
* non-traumatic
* minimally or non-invasive
* associated with a low incidence of adverse events such as dehiscence and infection
* yielding acceptable cosmetic results

ZipLine Medical, Inc. is a Campbell, California-based company that has developed a novel, non-invasive skin closure device called Zip Surgical Skin Closure to replace sutures, staples and glue for closure of the skin layer for surgical incisions or laceration repair. In the USA, the device has been classified by the FDA as a Class I, 510(k) Exempt device and began commercial use in the USA in April 2013.

The ZipLine Device has been clinically demonstrated benefits include (references included later in this document):

* Closure speed faster/superior to (and less variable compared to) sutures
* Suture-like cosmetic outcome
* Reduction in post-surgical care costs
* Fewer closure-related wound issues
* Greater patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age and older
2. Primary C-section
3. Patients willing and able to complete study protocol

Exclusion Criteria:

1. Known bleeding disorder not caused by medication
2. Known personal or family history of keloid formation or scar hypertrophy
3. Known allergy or hypersensitivity to non-latex skin adhesives
4. Atrophic skin deemed clinically prone to blistering
5. Any skin disorder affecting wound healing
6. Any other condition that in the opinion of the investigator would make a particular subject unsuitable for this study
7. Emergent C-Section
8. Non-primary C-Section

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Time of Procedure Closure | Procedure Closure - Zip or Suture touches skin until skin is closed
  Upon closure of the Cesarean incision - Zip or Suture touches skin to close incision
Cosmetic Visual Analogue Scale (CVAS) | 3 months
  100-mm Cosmetic Visual Analogue Scale (CVAS) for incision appearance

SECONDARY OUTCOMES:
Surgeon Closure Method Satisfaction | Procedure, 3-5 days, 3 months
  Satisfaction with closure method, scar appearance
Patient Closure Method Satisfaction | 3-5 days, 14 days, 3 months
  Satisfaction with closure method, scar appearance
Patient Pain and Discomfort by Subject Questionnaire | 3-5 days, 14 days, 3 months
  Pain associated with the closure method and level of discomfort during use will be asked by questionnaire
Incidence and severity of Adverse Events | Procedure, 3-5 days, 14 days, 3 months
  The incidence and severity of adverse events (AE) associated with Zip device and control will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Elias Castel, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No